CLINICAL TRIAL: NCT06397742
Title: Assessing the Implementation of Myofascial Techniques in Patients With Symptoms of Accessory Nerve Damage After Oncologic Treatment in the Head and Neck Regions
Brief Title: Assessing the Implementation of Myofascial Techniques in Patients With Accessory Nerve Damage After Oncologic Treatment
Acronym: PHYSIOACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Greater Poland Cancer Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHYSIOACCESS
Record Dates: First submitted 2024-04-15; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2020-03

CONDITIONS: Accessory Nerve Injuries; Physical Therapy
Keywords: head and neck cancer; nerve dysfunction; physical therapy
MeSH Terms: conditions — Accessory Nerve Injuries; Head and Neck Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study will recruit patients who underwent surgical therapy for head and neck cancer, with one-sided removal of lymph nodes, and who present symptoms of accessory nerve dysfunction. The group will be recruited from patients who underwent the surgical treatment in Greater Poland Cancer Centre. Outline of the two interventions will be presented to each patient, after which the patient will choose the preferred intervention.
  All patients from the study group were treated at the Head and Neck Surgery and Laryngological Oncology Clinic at the Poznań University of Medical Science.
  The study group comprised 9 women and 16 men with an average of 51.1 y.o., and the control group comprised 6 women and 17 men with an average of 50,8y.o.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity under supervision (Experimental): The subjects receive physical therapy three times a week for 45 minutes, during a six-week period under professional supervision.
  Interventions: Other: Physical therapy - myofascial techniques
- Home exercise (Active Comparator): The subjects receive a set of exercises and a recommendation to perform them at least three times a week for 45 minutes.
  To ensure compliance the subjects receive journals to record the performed exercises. Additionally subjects are contacted by phone to motivate them to exercise with adequate intensity. Furthermore the proper exercise technique is verified at periodic control visits.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — Patients received a set of exercises to execute at home. The home exercise program comprised 12 exercises conducted in sequence:
  1. Symmetrical shoulder raises with retraction
  2. Rolling upper extremities using a ball
  3. Symmetrical shoulder raises
  4. Band exercises strengthening the upper girdle and arm
  5. Exercise of the shoulder joint flexors
  6. Side arm raises in supine position
  7. Lateral arm raises in supine position
  8. Head raises with rotation in supine position
  9. Side arm raises in prone position
  10. Front arm raises in prone position
  11. Rising and lowering the upper girdle in prone position
  12. Neck muscles stretches
  Other Names: Home exercise program
  Arms: Home exercise
Other: Physical therapy - myofascial techniques — Physical therapy program comprised five parts. I. Fascial manipulation targeted three most active center of coordination - center of fusion points within head, neck, shoulder, shoulder blade, or chest - during each session, time depending on the patients' adaptability.
  II. Manual mobilization of the scar area with each training session including: active myofascial stretching; manual scar mobilization by stretching perpendicularly and in parallel with the scar; soft tissue mobilization by rolling and pulling the surface tissues; myofascial relaxation by breaking through restrictions.
  III. Relaxation of muscle contractures using post-isometric muscle relaxation of the scalene muscle, sternocleidomastoid muscle, and neck muscles - until the sessions provided no muscle elongation.
  IV. Neuromuscular stimulation with proprioceptive neuromuscular facilitation - included scapula movement patterns, dynamic reversal, stabilizing reversal, upper extremity movement patterns.
  Other Names: Physical therapy program
  Arms: Physical activity under supervision

SUMMARY:
The majority of head and neck cancers develop locally and regionally. Therefore, to reduce the risk of metastasis, 90% of surgeries performed in the head and neck area include the removal of regional lymph nodes and delivery of radiotherapy.

As a consequence of radical surgery affecting the lymphatic system in the neck area, there exists a risk of damage to the cervical plexus branch (C1-C4) or the accessory nerve. Patients with damage to this nerve develop disability involving limitations to the head flexion, extension, and rotation, asymmetric shoulder blades, disturbed shoulder joint abduction, flexion, and external rotation (supination). Additionally, patients often suffer from pain, numbness, swelling, and body asymmetry.

Subject literature does not describe in a detailed and comprehensive way the physiotherapeutic procedures to be applied in case of a damaged accessory nerve as a complication after cancer treatment. Unfortunately, it is often related to patients' limited access to an effective therapy. Available information on the rehabilitation procedures is limited and it mostly focuses on exercise recommendations. An analysis of the subject literature does not show any information on the efficiency of applying the myofascial techniques for treating deficiencies related to the damage of the accessory nerve.

In the current project the investigators plan to assess the effectiveness of a physical therapy intervention comprising myofascial techniques as compared to a set of exercises designed for performing individually in head and neck cancer patients with accessory nerve damage after surgical head and neck cancer treatment. The primary outcome will be physiotherapeutic procedures to be applied in case of a damaged accessory nerve as a complication after cancer treatment. The secondary outcomes will include the efficiency of applying the myofascial techniques for treating deficiencies related to the damage of the accessory nerve.

DETAILED DESCRIPTION:
The majority of head and neck cancers develop locally and regionally. Therefore, to reduce the risk of metastasis, 90% of surgeries performed in the head and neck area, include the removal of regional lymph nodes and delivery of radiotherapy.

As a consequence of radical surgery affecting the lymphatic system in the neck area, there exists a risk of damage to the cervical plexus branch (C1-C4) or the accessory nerve. However, depending on the cancer stage, in numerous cases it is possible to successfully save bodily structures and maintain continuation of nerves.

The analysis of complications shows that about 80% of patients communicate subjective discomforts of upper limb on the side of the surgery. After surgery treatment including lymphadenectomy (lymph node dissection) in the head and neck area, 60% of patients suffer from the damage or dysfunction of the accessory nerve.

As a consequence, there are numerous symptoms limiting the normal functioning of a patient. Among the most frequent symptoms of accessory nerve damage is a muscle dysfunction on the side of the nerve damage (trapezius muscle, sternocleidomastoid muscle). As a result of the accessory nerve damage, patients develop disability due to limitations to the head flexion, extension, and rotation, asymmetric shoulder blades, disturbed shoulder joint abduction, flexion, and external rotation (supination). Additionally, patients suffer from pain, numbness, swelling, and body asymmetry. Subject literature does not describe in a detailed and comprehensive way the physiotherapeutic procedures to be applied in case of a damaged accessory nerve as a complication after cancer treatment. Unfortunately, endurance of the impairment is often related to patients' limited access to an effective therapy

Purpose of the research:

The aim of this study is to assess the effectiveness of a physical therapy intervention comprising myofascial techniques as compared to a set of exercises designed for performing individually in head and neck cancer patients with accessory nerve dysfunction after surgical head and neck cancer treatment. The study will include patients treated surgically for head and neck cancer with one-sided lymphadenectomy in the head and neck region who present with pain, restricted mobility or muscle atrophy. Recruited patients will be divided into one of two groups: the first group will receive physical therapy including myofascial techniques performed by the physical therapist three times a week for 45 minutes, and the second group will receive a specially designed set of exercises to perform at home three times a week for 45 minutes. The intervention will last six weeks and patients will be assessed before and after intervention. Patient's neuromuscular condition will be examined using surface electromyography (sEMG), pain at rest, during shoulder flexion, and on trapezius muscle palpation will be measured using Visual Analogue Scale, and quality of life will be assessed using modified Neck Dissection Impairment Index (NDII) questionnaire.

Specific aims:

* To create an algorithm of physiotherapeutic procedures in case of the dysfunction of the accessory nerve and related complications.
* To assess the effect of applied techniques on the mobility of the cervical section of the spine.
* To assess the influence of the therapy on the mobility of the shoulder girdle on the post-surgery side.
* To assess the influence of the therapy on patients' pain related discomfort.
* To assess the feasibility of applying sEMG (surface electromyography) to verify the efficiency of the therapy.

ELIGIBILITY:
Inclusion Criteria:

* patients treated surgically for head and neck cancer with one-sided lymphadenectomy in the head and neck region,
* symptoms of damage to the accessory nerve,
* Eastern Cooperative Oncology Group (ECOG) scale 0-2,

Exclusion Criteria:

* local recurrence,
* distant metastases,
* cardiorespiratory failure,
* pain symptoms exceeding patients adaptability,
* decline of the patient's level of functioning to 3-4 in ECOG scale.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Shoulder range of motion: flexion, measured in degrees | within one week pre-intervention and one week after the intervention
  Shoulder range of motion: flexion, measured in degrees
Shoulder range of motion: abduction, measured in degrees | within one week pre-intervention and one week after the intervention
  Shoulder range of motion: abduction, measured in degrees
Shoulder range of motion: extension, measured in degrees | within one week pre-intervention and one week after the intervention
  Shoulder range of motion: extension, measured in degrees
Shoulder range of motion: rotation, measured in degrees | within one week pre-intervention and one week after the intervention
  Shoulder range of motion: rotation, measured in degrees

SECONDARY OUTCOMES:
Cervical spine range of motion: cervical flexion, measured in degrees | within one week pre-intervention and one week after the intervention
  Cervical spine range of motion: cervical flexion, measured in degrees
Cervical spine range of motion: cervical extension, measured in degrees | within one week pre-intervention and one week after the intervention
  Cervical spine range of motion: cervical extension, measured in degrees
Cervical spine range of motion: cervical lateral flexion, measured in centimetres | within one week pre-intervention and one week after the intervention
  Cervical spine range of motion: cervical lateral flexion, measured in centimetres
Cervical spine range of motion: cervical rotation, measured in centimetres | within one week pre-intervention and one week after the intervention
  Cervical spine range of motion: cervical rotation, measured in centimetres
Passive skeletal muscle tone | within one week pre-intervention and one week after the intervention
  Passive skeletal muscle tone in the upper trapezius on both sides, measured by surface electromyography (sEMG) amplitude
Skeletal muscle tone | within one week pre-intervention and one week after the intervention
  Skeletal muscle tone in the upper trapezius on both sides, measured at one second of muscle activation using sEMG amplitude
Skeletal muscle fatigue | within one week pre-intervention and one week after the intervention
  Skeletal muscle fatigue in the upper trapezius on both sides, measured as the difference between sEMG amplitude at one second and at the last second of muscle activation
Assessment of pain symptoms using Visual Analogue Scale (VAS) measured at rest, during shoulder flexion, and during trapezius muscle palpation; a single scale questionnaire, with range of points 1-10, with higher score meaning more intense pain | within one week pre-intervention and one week after the intervention
  Assessment of pain symptoms using Visual Analogue Scale (VAS) measured at rest, during shoulder flexion, and during trapezius muscle palpation; a single scale questionnaire, with range of points 1-10, with higher score meaning more intense pain
Quality of life after neck dissection, scored based on the Neck Dissection Impairment Index (NDII) questionnaire, a single scale with range of points 5-50, with a higher score meaning worse quality of life | within one week pre-intervention and one week after the intervention
  Quality of life after neck dissection, scored based on the Neck Dissection Impairment Index (NDII) questionnaire, a single scale with range of points 5-50, with a higher score meaning worse quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Górecki, PhD, Principal Investigator — Greater Poland Cancer Centre
Locations (1):
- Ewa Tanska, Poznan, Polska, Poland

REFERENCES:
- [Background] Bhattacharyya N. The increasing workload in head and neck surgery: An epidemiologic analysis. Laryngoscope. 2011 Jan;121(1):111-5. doi: 10.1002/lary.21193. PMID 21154824
- [Background] Popovski V, Benedetti A, Popovic-Monevska D, Grcev A, Stamatoski A, Zhivadinovik J. Spinal accessory nerve preservation in modified neck dissections: surgical and functional outcomes. Acta Otorhinolaryngol Ital. 2017 Oct;37(5):368-374. doi: 10.14639/0392-100X-844. PMID 29165431
- [Background] Marszałek W.S., Majchrzycki M., Golusiński W.: Dysfunctions of the locomotor system. Physiotherapy in head and neck cancer. Poznan: Poznan University of Medical Sciences Publishing House, 2012, ISBN: 978-83-7597-161-3
- [Background] Guru K, Manoor UK, Supe SS. A comprehensive review of head and neck cancer rehabilitation: physical therapy perspectives. Indian J Palliat Care. 2012 May;18(2):87-97. doi: 10.4103/0973-1075.100820. PMID 23093823
- [Background] Goldstein DP, Ringash J, Bissada E, Jaquet Y, Irish J, Chepeha D, Davis AM. Scoping review of the literature on shoulder impairments and disability after neck dissection. Head Neck. 2014 Feb;36(2):299-308. doi: 10.1002/hed.23243. Epub 2013 Apr 1. PMID 23554002
- [Background] Dijkstra PU, van Wilgen PC, Buijs RP, Brendeke W, de Goede CJ, Kerst A, Koolstra M, Marinus J, Schoppink EM, Stuiver MM, van de Velde CF, Roodenburg JL. Incidence of shoulder pain after neck dissection: a clinical explorative study for risk factors. Head Neck. 2001 Nov;23(11):947-53. doi: 10.1002/hed.1137. PMID 11754498
- [Background] Koybasioglu A, Bora Tokcaer A, Inal E, Uslu S, Kocak T, Ural A. Accessory nerve function in lateral selective neck dissection with undissected level IIb. ORL J Otorhinolaryngol Relat Spec. 2006;68(2):88-92. doi: 10.1159/000091209. Epub 2006 Jan 27. PMID 16446553
- [Background] Carvalho AP, Vital FM, Soares BG. Exercise interventions for shoulder dysfunction in patients treated for head and neck cancer. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD008693. doi: 10.1002/14651858.CD008693.pub2. PMID 22513964
- [Background] Day JA, Stecco C, Stecco A. Application of Fascial Manipulation technique in chronic shoulder pain--anatomical basis and clinical implications. J Bodyw Mov Ther. 2009 Apr;13(2):128-35. doi: 10.1016/j.jbmt.2008.04.044. Epub 2008 Jun 24. PMID 19329049
- [Background] Laska T, Hannig K. Physical therapy for spinal accessory nerve injury complicated by adhesive capsulitis. Phys Ther. 2001 Mar;81(3):936-44. PMID 11268158
- [Background] McGarvey AC, Osmotherly PG, Hoffman GR, Chiarelli PE. Impact of neck dissection on scapular muscle function: a case-controlled electromyographic study. Arch Phys Med Rehabil. 2013 Jan;94(1):113-9. doi: 10.1016/j.apmr.2012.07.017. Epub 2012 Aug 1. PMID 22864015
- [Background] McGarvey AC, Hoffman GR, Osmotherly PG, Chiarelli PE. Maximizing shoulder function after accessory nerve injury and neck dissection surgery: A multicenter randomized controlled trial. Head Neck. 2015 Jul;37(7):1022-31. doi: 10.1002/hed.23712. Epub 2014 Jul 11. PMID 25042422
- [Background] Hindle KB, Whitcomb TJ, Briggs WO, Hong J. Proprioceptive Neuromuscular Facilitation (PNF): Its Mechanisms and Effects on Range of Motion and Muscular Function. J Hum Kinet. 2012 Mar;31:105-13. doi: 10.2478/v10078-012-0011-y. Epub 2012 Apr 3. PMID 23487249
- [Background] Gane EM, McPhail SM, Hatton AL, Panizza BJ, O'Leary SP. The relationship between physical impairments, quality of life and disability of the neck and upper limb in patients following neck dissection. J Cancer Surviv. 2018 Oct;12(5):619-631. doi: 10.1007/s11764-018-0697-5. Epub 2018 May 16. PMID 29770954
- [Background] Tarkan Ö., Tuncer Ü., Bozdemir H., Sarpel T., Özdemir S., Surmelioglu Ö.: Clinical and electrophysiological evaluation of shoulder functions in spinal accessory nerve-preserving neck dissection. Turk J Med Sci, 2012; 42(5): 852-860